CLINICAL TRIAL: NCT03696511
Title: Multicentric Clinical Study Protocol on Primary Stability of STORM® Miniscrew
Brief Title: Miniscrews Primary Stability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Genova (Other)
Collaborators: Università degli Studi di Brescia (Other); Alfonso X El Sabio University (Other)
Responsible Party: Principal Investigator, Marco Migliorati, Lecturer, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE-BS-MA MRCT
Record Dates: First submitted 2018-07-18; First posted 2018-10-04 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2018-10

CONDITIONS: Orthodontic Appliance Complication
Keywords: Miniscrew

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: data sheet will be blinded for the analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1:maxillary insertion (Active Comparator): Orthodontic miniscrew insertion; maxillary insertion. buccal
  Interventions: Device: Orthodontic miniscrew insertion
- group 2: mandible insertion (Active Comparator): Orthodontic miniscrew insertion; mandible insertion.
  Interventions: Device: Orthodontic miniscrew insertion
- group 3: palatal insertion (Active Comparator): Orthodontic miniscrew insertion; palatal insertion
  Interventions: Device: Orthodontic miniscrew insertion

INTERVENTIONS:
Device: Orthodontic miniscrew insertion — orthodontic treatment using miniscrews as anchorage reinforcement

SUMMARY:
Orthodontic Miniscrew primary stability is essential for success and long term results.

The aim of the present study is to evaluate Bone Properties and Torque insertion values and how they could be related to primary stability and success rate of miniscrew.

DETAILED DESCRIPTION:
Orthodontic miniscrews are intraoral anchorage devices designed to support biomechanics during orthodontic tooth movement. Also known as miniscrews, mini-implants, microscrews, or temporary anchorage devices, they are made of a head, a neck, and a threaded shank. The head may show different designs (bracket-like, rounded with slot, etc.) the threaded shank is generally cylindrical, tapered or a combination of the two, and may be self-tapping (i.e. requiring a pre-drilled pilot hole) and/or self-drilling (not requiring a pilot hole). Because of their small diameter, they may be implanted in a wide variety of anatomic sites, such as the alveolar interradicular spaces or the palatal cortical bone, in order to attend to treatment anchorage needs. The loading protocol for miniscrews loading can be as immediate as delayed; in the beginning in literature was indicated a non-specific period of healing and osseointegration before a screw inserted in the mandible could be loaded; the importance of a healing period was derived by several studies on Branemark protocol on implants. Further experimental studies on orthodontic load were not able to demonstrate loaded implant loosening, even when loads were applied immediately, so that an immediate loading protocol for orthodontic miniscrews appeared as reasonable. Costa and Melsen studied the tissue reaction around the immediately loaded screws in an animal model and suggested the use of immediately loaded screws as an intra-oral extra-dental anchorage. Histomorphometric analyses have shown that the immediate loading of miniscrew implants may help to activate bone remodeling and increase the mineral contents at the loaded region. Compared to traditional endosseous implants, orthodontic miniscrews have relatively high failure rates, varying from 16.4% to 39% ; according to recent reviews, the average failure rate is believed to be less than 20%. Many factors have been proposed to be associated to success rate; among these age, gender, jaw (maxilla or mandible), placement site, tissue mobility (firm or movable tissue), inflammation, distance to the root, insertion torque, loading time, type, length, and diameter of the miniscrew. Recently, an experimental study on primary stability found that bone properties are more important than the screw geometry in establishing primary mechanical retention. Thus the aim of this study is to deeply analyze the bone role related to the success of miniscrews analyzing both insertion/removal torque values, both bone characteristics by the mean of x-rays.

ELIGIBILITY:
Inclusion Criteria:

* patient who need ortho treatment with miniscrew
* permanent dentition

Exclusion Criteria:

* bone pathologies
* systemic disease

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Success | From the moment the screw will be placed, measuring maximum insertion torque, through study completion, when the screws will be removed, measuring removal torque. An average duration of screw of 10-12 months is expected.
  How many screws don't fail. Success if the screw remain stable until the end of biomechanics applied.

SECONDARY OUTCOMES:
MIT | The date when, for each patient, the miniscrew will be inserted. Registered as the insertion date (day). Up to 12 months from orthodontic therapy beginning. The event is determined from date of randomization list creation until the day of screw insertion
  miniscrew maximum insertion torque: The moment when the screw will be placed, the maximum insertion torque will be registered at the insertion time, with a analogical screwdriver, measured in Ncm
MRT | The date when, for each patient,the miniscrew will be removed.Registered as the removal date (day).Up to 24 months after miniscrew insertion.The event is determined from date of randomization list creation until the day of screw removal, up to 48 months
  maximum removal torque. Maximum removal torque will be recorded using an analogical screwdriver at the completion of screw insertion. MRT is a unique value expressed in Ncm measured when the screws will be removed.

OTHER OUTCOMES:
Cortical thickness | At the beginning of the orthodontic treatment, before any dental movement occurred. Time frame is from randomization list and beginning of orthodontic treatment, up to 24 months.
  cortical thickness measured in mm, a. Both values will be evaluated on CBCT images acquired before orthodontic treatment beginning
Marrow bone density | At the beginning of the orthodontic treatment, before any dental movement occurred. Time frame is from randomization list and beginning of orthodontic treatment, up to 24 months.
  marrow/cortical bone density measured with HU values. Images will be evaluated with dedicated software for image analysis

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Orthodontic Departments, Brescia
  - Orthodontic Department, Genova
- Universidad Alfonso X El Sabio (UAX), Madrid, Spain

REFERENCES:
- [Result] Migliorati M, Drago S, Dalessandri D, Lagazzo A, Gallo F, Capurro M, Silvestrini-Biavati A. On the stability efficiency of anchorage self-tapping screws: Ex vivo experiments on miniscrew implants used in orthodontics. J Mech Behav Biomed Mater. 2018 May;81:46-51. doi: 10.1016/j.jmbbm.2018.02.019. Epub 2018 Feb 19. PMID 29482179
- [Result] Watanabe T, Miyazawa K, Fujiwara T, Kawaguchi M, Tabuchi M, Goto S. Insertion torque and Periotest values are important factors predicting outcome after orthodontic miniscrew placement. Am J Orthod Dentofacial Orthop. 2017 Oct;152(4):483-488. doi: 10.1016/j.ajodo.2017.01.026. PMID 28962732
- [Result] Inoue M, Kuroda S, Yasue A, Horiuchi S, Kyung HM, Tanaka E. Torque ratio as a predictable factor on primary stability of orthodontic miniscrew implants. Implant Dent. 2014 Oct;23(5):576-81. doi: 10.1097/ID.0000000000000138. PMID 25192157
- [Result] Watanabe H, Deguchi T, Hasegawa M, Ito M, Kim S, Takano-Yamamoto T. Orthodontic miniscrew failure rate and root proximity, insertion angle, bone contact length, and bone density. Orthod Craniofac Res. 2013 Feb;16(1):44-55. doi: 10.1111/ocr.12003. Epub 2012 Sep 3. PMID 23311659
- [Result] Migliorati M, Drago S, Gallo F, Amorfini L, Dalessandri D, Calzolari C, Benedicenti S, Silvestrini-Biavati A. Immediate versus delayed loading: comparison of primary stability loss after miniscrew placement in orthodontic patients-a single-centre blinded randomized clinical trial. Eur J Orthod. 2016 Dec;38(6):652-659. doi: 10.1093/ejo/cjv095. Epub 2016 Jan 4. PMID 26728036